CLINICAL TRIAL: NCT05949749
Title: A Retrospective Study Reveals the Relationship Between gp42-IgG Epitopes and EBV-associated NPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-631-01
Record Dates: First submitted 2023-06-21; First posted 2023-07-18 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case
  Interventions: Diagnostic Test: Epitope exploration
- Control
  Interventions: Diagnostic Test: Epitope exploration

INTERVENTIONS:
Diagnostic Test: Epitope exploration — Explore the epitope landscape of gp42-IgG of cases in comparison with that of controls.

SUMMARY:
Epstein-barr virus (EBV) infection is a necessary factor of nasopharyngeal carcinoma (NPC). The incidence of NPC in endemic regions reaches 24.60/100,000 people, far higher than that of the worldwide average. However, no EBV prophylactic vaccines is clinically available so far, which is largely hampered by the difficulties in selecting optimal vaccine design target out of 13 glycoproteins on the surface of EBV. In this study, we utilized humanized gp42-IgG antibodies to explore the dominant epitopes of gp42, one of the functional EBV glycoproteins during virus entry, to facilitate prophylactic vaccine design.

ELIGIBILITY:
Inclusion Criteria:

* Controls underwent physical examinations or primary NPC cases confirmed by pathology or cytology.
* If cases, at stage I-IVB diagnosed by radiology according to AJCC/UICC 8th.
* If cases, Karnofsky score (KFS)≥70, estimated survival span>12 months.
* If cases, no disordered of major organs is found; blood test, liver, and kidney functions are basically normal.
* If cases, at least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.

Exclusion Criteria:

* History of other malignant diseases.
* History of severe systemic diseases or heart, lung, liver, or kidney disfunction.
* History of severe neurological, metal, endocrine diseases.
* History of HBV, HCV, HIV, TP, or TB infection.
* If controls, physical examination reveals systemic diseases including malignant diseases.
* If cases, incomplete blood and pathological sample data.
* If cases, not receiving primary treatment in this facility.
* Other individuals investigators find not suitable for the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chinese.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Dominant gp42-IgG epitopes in cases | Baseline
  Dominant gp42-IgG epitopes revealed by ELISA with non-competitive monoclonal humanized antibodies against gp42 will be compared between cases and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ming Huang, M.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided